CLINICAL TRIAL: NCT02705768
Title: Effect of Carbamazepine and Oxcarbazepine on Serum Neuron-specific Enolase and S100B in Focal Seizures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, RITUPARNA MAITI, Associate Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T/IM -NF/Pharm/15/30
Record Dates: First submitted 2016-03-03; First posted 2016-03-11 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Seizures, Focal
Keywords: Neuron-specific enolase (NSE); Carbamazepine; Oxcarbazepine
MeSH Terms: conditions — Seizures | interventions — Carbamazepine; Oxcarbazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy control (No Intervention): Twenty five (25) healthy individuals of same age group will serve as the control group. Control subjects will be evaluated at baseline only.
- Carbamazepine group (Experimental): Twenty five (25) patients recruited in this group will receive Tab. Carbamazepine. Carbamazepine will be started with a dose of 200 mg/day for one week and then increased to 400 mg/day for one week and then 600mg/day for next two weeks.
  Interventions: Drug: Carbamazepine
- Oxcarbazepine group (Experimental): Twenty five (25) patients recruited in this group will receive Tab. Oxcarbazepine. Oxcarbazepine will be started with 10mg/kg daily dose for one week followed by 15mg/kg daily for next one week and then will be increased to 20mg/kg for next two weeks.
  Interventions: Drug: Oxcarbazepine

INTERVENTIONS:
Drug: Carbamazepine — Carbamazepine will be started with a dose of 200 mg/day for one week and then increased to 400 mg/day for one week and then 600mg/day for next two weeks.
  Other Names: Tegretol
  Arms: Carbamazepine group
Drug: Oxcarbazepine — Oxcarbazepine will be started with 10mg/kg daily dose for one week followed by 15mg/kg daily for next one week and then will be increased to 20mg/kg for next two weeks.
  Other Names: Oxetol
  Arms: Oxcarbazepine group

SUMMARY:
The present study has been planned to assess the level of serum neuron-specific enolase (NSE) in focal seizures and its changes after antiepileptic therapy.

DETAILED DESCRIPTION:
Epileptic seizures can cause neuronal cell death, enhanced neurogenesis, axonal sprouting, dendritic changes, and reactive gliosis. Histopathological analyses have suggested that the initial insult and recurrent seizures contribute to the neuronal damage. Activation of mesial temporal structures is more likely to cause damage than that of other areas of brain; therefore, one of the consequences of prolonged seizures is selective neuronal loss in the hippocampus. The excitotoxic damage is considered the most important mechanism of injury but there is also evidence that programmed cell death contributes to neuronal damage.

Various biomarkers of brain damage have been studied in the context of epilepsy and brain damage but most widely investigated biochemical biomarker is neuron-specific enolase (NSE). NSE is γγ-isoenzyme of enolase involved in glycolysis pathway. NSE originates predominantly from the cytoplasm of neurons and neuroendocrine cells. Neuronal damage and impairment of blood brain barrier integrity can be detected by the release of NSE into cerebrospinal fluid (CSF) and eventually into blood. NSE is therefore regarded as a marker of neuronal damage and prognosis in various disorders associated with cell damage in the central or peripheral nervous system.

CSF and serum NSE levels obtained within first 48 hours were found to be elevated and correlated well with the duration of epilepsy and outcome of patients. Some studies have shown elevated NSE levels in temporal lobe epilepsy, after single tonic-clonic seizures, and status epilepticus. Literature review reveals that there is lack of data on serum NSE in focal seizures and there is no study on the effect of antiepileptic drugs on the level of serum NSE. So the present study has been planned to assess the level of serum NSE in focal seizures and its changes after antiepileptic therapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients with the clinical diagnosis of localization related epilepsy/focal seizure (International League Against Epilepsy 2010) with a history of an episode of seizure within 48 hours of presentation
* Treatment naïve patients or patients who had not taken any treatment for at least 3 weeks before inclusion.

Exclusion Criteria:

* History of any recent traumatic brain injury, cerebral ischemia/transient ischemic attack/stroke
* Patients with neuroendocrinal tumours
* History of any invasive neurosurgical /non-invasive neuropsychiatric procedure.
* Patients who are already under treatment for the presenting conditions.
* Medication history of psychoactive or central nervous system depressant drugs
* Pregnant and nursing women

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Serum neuron-specific enolase (NSE) and S100B | Change from baseline over 4 weeks
  Method: ELISA

SECONDARY OUTCOMES:
Severity of seizure episode as measured by Chalfont-National Hospital seizure severity scale (NHS3) | Change from baseline over 4 weeks
  The scale was developed at the Chalfont Centre for Epilepsy based on the Chalfont Seizure Severity Scale. It can be used to measure the severity of the seizures and to evaluate anti-epileptic agents during clinical trials.
Quality of life as assessed by Quality of Life in Epilepsy Inventory (QOLIE-31) | Change from baseline over 4 weeks
  Quality of Life in Epilepsy Inventory (QOLIE-31) contains seven multi-item scales that tap the following health concepts: emotional well-being, social functioning, energy/fatigue, cognitive functioning, seizure worry, medication effects, and overall quality of life. A QOLIE31 overall score is obtained using a weighted average of the multi-item scale scores.

CONTACTS AND LOCATIONS:
Overall Officials: DEBASISH HOTA, DM, Study Director — AIIMS, Bhubaneswar
Locations (1):
- AIIMS, Bhubaneswar, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sutula TP. Mechanisms of epilepsy progression: current theories and perspectives from neuroplasticity in adulthood and development. Epilepsy Res. 2004 Jul-Aug;60(2-3):161-71. doi: 10.1016/j.eplepsyres.2004.07.001. PMID 15380560
- [Result] Holmes GL. Seizure-induced neuronal injury: animal data. Neurology. 2002 Nov 12;59(9 Suppl 5):S3-6. doi: 10.1212/wnl.59.9_suppl_5.s3. PMID 12428025
- [Result] Henshall DC, Clark RS, Adelson PD, Chen M, Watkins SC, Simon RP. Alterations in bcl-2 and caspase gene family protein expression in human temporal lobe epilepsy. Neurology. 2000 Jul 25;55(2):250-7. doi: 10.1212/wnl.55.2.250. PMID 10908900
- [Result] Kato K, Ishiguro Y, Suzuki F, Ito A, Semba R. Distribution of nervous system-specific forms of enolase in peripheral tissues. Brain Res. 1982 Apr 15;237(2):441-8. doi: 10.1016/0006-8993(82)90455-3. PMID 7044473
- [Result] Royds JA, Davies-Jones GA, Lewtas NA, Timperley WR, Taylor CB. Enolase isoenzymes in the cerebrospinal fluid of patients with diseases of the nervous system. J Neurol Neurosurg Psychiatry. 1983 Nov;46(11):1031-6. doi: 10.1136/jnnp.46.11.1031. PMID 6317805
- [Result] DeGiorgio CM, Correale JD, Gott PS, Ginsburg DL, Bracht KA, Smith T, Boutros R, Loskota WJ, Rabinowicz AL. Serum neuron-specific enolase in human status epilepticus. Neurology. 1995 Jun;45(6):1134-7. doi: 10.1212/wnl.45.6.1134. PMID 7783877
- [Result] Correale J, Rabinowicz AL, Heck CN, Smith TD, Loskota WJ, DeGiorgio CM. Status epilepticus increases CSF levels of neuron-specific enolase and alters the blood-brain barrier. Neurology. 1998 May;50(5):1388-91. doi: 10.1212/wnl.50.5.1388. PMID 9595992
- [Result] Palmio J, Keranen T, Alapirtti T, Hulkkonen J, Makinen R, Holm P, Suhonen J, Peltola J. Elevated serum neuron-specific enolase in patients with temporal lobe epilepsy: a video-EEG study. Epilepsy Res. 2008 Oct;81(2-3):155-60. doi: 10.1016/j.eplepsyres.2008.05.006. Epub 2008 Jul 1. PMID 18595663
- [Result] Chang CC, Lui CC, Lee CC, Chen SD, Chang WN, Lu CH, Chen NC, Chang AY, Chan SH, Chuang YC. Clinical significance of serological biomarkers and neuropsychological performances in patients with temporal lobe epilepsy. BMC Neurol. 2012 Mar 14;12:15. doi: 10.1186/1471-2377-12-15. PMID 22417223
- [Result] Buttner T, Lack B, Jager M, Wunsche W, Kuhn W, Muller T, Przuntek H, Postert T. Serum levels of neuron-specific enolase and s-100 protein after single tonic-clonic seizures. J Neurol. 1999 Jun;246(6):459-61. doi: 10.1007/s004150050383. PMID 10431771
- [Result] Rabinowicz AL, Correale J, Boutros RB, Couldwell WT, Henderson CW, DeGiorgio CM. Neuron-specific enolase is increased after single seizures during inpatient video/EEG monitoring. Epilepsia. 1996 Feb;37(2):122-5. doi: 10.1111/j.1528-1157.1996.tb00002.x. PMID 8635421
- [Result] Duncan JS, Sander JW. The Chalfont Seizure Severity Scale. J Neurol Neurosurg Psychiatry. 1991 Oct;54(10):873-6. doi: 10.1136/jnnp.54.10.873. PMID 1744641
- [Result] Cramer JA, French J. Quantitative assessment of seizure severity for clinical trials: a review of approaches to seizure components. Epilepsia. 2001 Jan;42(1):119-29. doi: 10.1046/j.1528-1157.2001.19400.x. PMID 11207795
- [Result] Cramer JA, Perrine K, Devinsky O, Bryant-Comstock L, Meador K, Hermann B. Development and cross-cultural translations of a 31-item quality of life in epilepsy inventory. Epilepsia. 1998 Jan;39(1):81-8. doi: 10.1111/j.1528-1157.1998.tb01278.x. PMID 9578017
- [Derived] Maiti R, Mishra BR, Sanyal S, Mohapatra D, Parida S, Mishra A. Effect of carbamazepine and oxcarbazepine on serum neuron-specific enolase in focal seizures: A randomized controlled trial. Epilepsy Res. 2017 Dec;138:5-10. doi: 10.1016/j.eplepsyres.2017.10.003. Epub 2017 Oct 6. PMID 29028517